CLINICAL TRIAL: NCT05008445
Title: A Phase I/II, Open-Label, Multiple Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM-102 Monotherapy or Combination Therapy in Patients With CLDN18.2-Positive Advanced Solid Tumors
Brief Title: Study of LM-102 in Patients With Advance Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company adjusted strategy
Sponsor: LaNova Medicines Development Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM102-01-102
Record Dates: First submitted 2021-07-27; First posted 2021-08-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- LM-102 Dose Escalation Level 1, 3mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  first dose: 3mg/kg, Q3W;
  Interventions: Biological: LM-102 Injection
- LM-102 Dose Escalation Level 2, 10mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  Second dose: 10mg/kg, Q3W;
  Interventions: Biological: LM-102 Injection
- LM-102 Dose Escalation Level 3, 20mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  Third dose: 20mg/kg, Q3W;
  Interventions: Biological: LM-102 Injection
- LM-102 Dose Escalation Level 4, 30mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  Four dose: 30mg/kg, Q3W;
  Interventions: Biological: LM-102 Injection
- LM-102 Dose Escalation Level 5, 40mg/kg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  Five dose: 40mg/kg, Q3W;
  Interventions: Biological: LM-102 Injection
- LM-102 (RP2D-1) combined with SOC Dose Escalation (Experimental): During the dose escalation of LM-102 combined with SOC,the next lower dose groups (RP2D-1) of LM-102 monotherapy's RP2D will be adopted as the starting dose.
  Interventions: Combination Product: LM-102 Injection combined with SOC
- LM-102 (RP2D) combined with SOC Dose Escalation (Experimental): During the dose escalation of LM-102 combined with SOC,(If applicable) LM-102 monotherapy's RP2D will be adopted as the starting dose.
  Interventions: Combination Product: LM-102 Injection combined with SOC

INTERVENTIONS:
Biological: LM-102 Injection — LM-102 Injection with dose escalation stage of 3mg/kg up to 40mg/kg, as well as dose expansion stage with recommended dose level from dose escalation stage.
  Arms: LM-102 Dose Escalation Level 1, 3mg/kg; LM-102 Dose Escalation Level 2, 10mg/kg; LM-102 Dose Escalation Level 3, 20mg/kg; LM-102 Dose Escalation Level 4, 30mg/kg; LM-102 Dose Escalation Level 5, 40mg/kg
Combination Product: LM-102 Injection combined with SOC — LM-102 Injection with appropriate dose level(s), combined with SOC.
  Arms: LM-102 (RP2D) combined with SOC Dose Escalation; LM-102 (RP2D-1) combined with SOC Dose Escalation

SUMMARY:
This is an open label Phase I/II trial of LM-102 injection, a recombinant humanized monoclonal antibody targeting Claudin 18.2 (CLDN18.2). It is being tested in advanced solid tumors including gastric cancer/gastroesophageal junction adenocarcinoma, Pancreatic Cancer, Biliary Tract Cancer, esophageal adenocarcinoma and ovarian mucous carcinoma.

DETAILED DESCRIPTION:
This study includes phase I dose escalation and phase II dose expansion.

Phase I dose escalation consists of LM-102 monotherapy dose escalation (Part Ia) and LM-102 combination dose escalation (Part Ib):

Part Ia is LM-102 monotherapy dose escalation, will be conducted among the subjects with recurrent or refractory advanced solid tumors to determine the RP2D of LM-102 monotherapy;Statistical designs include an initial accelerated titration at the first dose level followed by the i3+3 design at other four dose levels ; Part Ib is the dose escalation of LM-102 combined with SOC, will be conducted in the subjects with advanced gastric and gastroesophageal junction adenocarcinoma(GC/GEJ), pancreatic cancer (PC)and biliary tract carcinoma(BTC), respectively in first setting or second setting, to explore the recommended dose of LM-102 in combination SOC for dose expansion, 4 cohorts are planned;

Phase II dose expansion consists of LM-102 monotherapy dose escalation (Part IIa) and LM-102 combination dose escalation (Part IIb):

Part IIa is the dose expansion of LM-102 monotherapy, 3 cohorts are planned in the subjects with CLDN18.2 positive, recurrent or refractory advanced GC/GEJ , PC , BTC , to explore the preliminary efficacy of LM-102 monotherapy in the target tumor types； Part IIb is the dose expansion of LM-102 in combination with SOC, 4 cohorts are planned in the subjects with advanced, CLDN18.2 positive, treatment naïve GC/GEJ, PC, BTC, and in the subjects with GC/GEJ who have progressed on first line treatment, with the aim to to explore the preliminary efficacy of LM-102 monotherapy in the target tumor types;

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled into the study only if they meet all of the following inclusion criteria:

1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent document prior to any procedure;
2. Aged between 18 to 75 years old, male or female when sign the Informed consent form (ICF);
3. Subjects who meet the criteria:

   Phase I dose escalation:

   Part Ia: Subjects have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and are intolerable for available standard therapy, or there is no available standard therapy.

   Part Ib:Subjects have been histologically or cytologically confirmed advanced solid tumors and meet the criteria as follows: No previous systemic chemotherapy was given for the recurrent or metastatic disease or for the subjects who have received curative treatment (including neo-adjuvant or adjuvant chemotherapy /radiotherapy, etc.), the interval between recurrence and the last dose of previous anti-cancer treatment must be more than 6 months.

   Phase II dose expansion: subjects with positive CLDN18.2 confirmed by central immunohistochemistry (IHC).

   Part IIa: Subjects have histological or cytological confirmation of recurrent or refractory advanced solid tumors, and are intolerable for available standard therapy, or there is no available standard therapy.

   Part IIb: Subjects have histological or cytological confirmation of advanced solid tumors and meet the criteria as follows: No previous systemic chemotherapy was given for the recurrent or metastatic disease, or for the subjects who have received curative treatment (including neo-adjuvant or adjuvant chemotherapy /radiotherapy, etc.), the interval between recurrence and the last dose of previous anti-cancer treatment must be more than 6 months;
4. At least one evaluable lesion for phase I and one measurable lesion for phase II according to RECIST v1.1;
5. ECOG score 0-1;
6. Life expectancy ≥ 3 months;
7. Subjects must have the following organ and marrow function in laboratory tests within 7 days prior to the first dose;
8. Subjects who are able to well communicate with investigators as well as understand and adhere to the requirements of this study.

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any of the following criteria:

1. Child-bearing potential female who have positive results in pregnancy test or are lactating;
2. Subjects who known to be allergic to the similar products or any of its excipients;
3. Exposure to any IMP, or participate in any other clinical trial within 21 days prior to 1st dosing of LM-102;
4. Subjects with anti-tumor treatment within 28 days prior to 1st dosing of LM-302, including radiotherapy, chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc.
5. Subjects who have received surgical or interventional treatment within 28 days prior to 1st dosing LM-102, with the exception for tumor biopsy, puncture, etc.;
6. Subjects who have received the treatment targeting to CLDN18.2 or ADCs;
7. Use of any live vaccines (e.g., against infectious diseases such as influenza, varicella etc.) within 28 days prior to 1st dosing of LM-102;
8. Subjects with the history of interstitial lung disease or drug-induced interstitial lung disease/pneumonitis;
9. Subjects who are taking therapeutic doses of anticoagulants such as heparin or vitamin K antagonists (except for preventive treatment at a stable dose);
10. Subjects with gastric outlet obstruction, persistent recurrent vomiting or uncontrolled/severe gastrointestinal hemorrhage, or ulcer within 28 days prior to 1st dosing;
11. Subjects who are unable to take the oral drugs, have the conditions that severely affect gastrointestinal absorption;
12. Subjects with known central nervous system (CNS) or meningeal metastasis;
13. Subjects who have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures;
14. Subjects who have severe cardiovascular disease;
15. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0;
16. Subjects with uncontrolled tumor-related pain.
17. Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection requiring antibiotics administration;
18. Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
19. HIV infection, active HBV and HCV infection;
20. Men and women who are unwilling to use appropriate contraceptive methods throughout the study period and for at least 6 months after the last use of LM-102;
21. Subjects who have psychiatric illness or social situations that would preclude study compliance;
22. Subjects who have another active malignancy which is likely to require treatment, and have the history of another malignancy within 2 years before the first dosing;
23. Subject who is determined as not eligible to participate in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence and case number of DLT (Dose Limiting Toxicity) during observation period | up to 21 days following first dose
  DLT is short for Dose Limiting Toxicity. dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Participant Safety as characterized by frequency and severity of adverse events(according to NCI CTCAE 5.0) | up to 31 days following last dose or other anti-cancer therapy
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Recommended Phase II Dose (RP2D) | up to 21 days following first dose
  The RP2D will be determined during the dose expansion stage of the study. RP2D will be determined using available safety and efficacy data.
Maximum Tolerated Dose (MTD） | up to 21 days following first dose
  The MTD is defined as the dose of which the toxicity rate is lower than the upper bound of EI p_T+ϵ_1= 0.35 and closest to the target toxicity rate of p_T= 0.3 during the DLT observation period (21 days after the first administration in cycle 1 on day 1).

SECONDARY OUTCOMES:
Area under plasma concentration vs time curve (AUC) for LM-102 | Up to finished circle 5 (each cycle is 21 days)
  changes in AUC over time in participants with LM-102
Peak plasma concentration (Cmax) for LM-102 | Up to finished circle 5 (each cycle is 21 days)
  Cmax is the maximum plasma concentration.
Time to maximum observed plasma concentration (Tmax) | Up to finished circle 5 (each cycle is 21 days)
  Tmax is the time in hrs/days it takes to reach Cmax after dosing with LM-102
Terminal elimination half life (t1/2) | Up to finished circle 5 (each cycle is 21 days)
  Time for the plasma level of LM-102 to decrease by 1/2 during the terminal elimination phase
Immunogenicity | up to 31 days following last dose
  by measurement of Incidence of anti-drug antibodies (ADA)
Disease Control Rate(DCR ) | through study completion, an average of 8 months.
  as measured by RECIST v1.1
Duration of Response (DOR) | through study completion, an average of 8 months.
  as measured by RECIST v1.1
Progression free survival (PFS) | through study completion, an average of 8 months.
  as measured by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Fudan Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No